CLINICAL TRIAL: NCT06442358
Title: BPP for ME: Self Biophysical Profile Proof of Concept
Brief Title: Self Biophysical Profile Using a Home Ultrasound Device Proof of Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseNmore (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00244136
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Perinatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm home ultrasound in pregnant women require BPP (Other): Pregnant participants will use Pulsenmore ES device to perform BPP while guided remotely by a clinician
  Interventions: Device: Pulsenmore ES home ultrasound device

INTERVENTIONS:
Device: Pulsenmore ES home ultrasound device — Pulsenmore ES device is a portable home used ultrasound device which allow the patient to perform an ultrasound scan from the comfort of their home under the supervision of a healthcare provider

SUMMARY:
The objective of this study is to assess if patients presenting for antenatal testing can complete a Bio Physical Score (BPP) with a home-use ultrasound with remote clinician guidance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Singleton pregnancy
* Gestational age ≥ 24 0/7 weeks
* No known major fetal or genetic anomalies (may include: isolated pyelectasis, isolated --VSD, multicystic dysplastic kidney, cleft lip/palate, club foot, etc.)
* Ability to understand and sign informed consent in English
* Ability to read and understand instructions in English
* Ability to hold an ultrasound probe and respond to clinician instructions
* BMI less than 40 at initial prenatal visit
* Scheduled biophysical profile (BPP)
* Any maternal/pregnancy complications requiring antenatal testing, including but not limited to intrauterine growth restriction, chronic or gestational hypertension, preexisting or gestational diabetes, autoimmune disorder, etc.

Exclusion Criteria:

* Multiple gestation
* Known major fetal structural anomaly or aneuploidy
* Known fetal or genetic anomalies
* Ruptured membranes
* Uterine complaints, such as painful contractions
* Maternal concern for decreased fetal movement
* Not evaluated vaginal bleeding (not including spotting)
* Fetal or maternal criteria that require urgent delivery
* BMI ≥ 40 at initial prenatal visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Assess feasibility and proof of concept that the Pulsenmore home ultrasound device can be used to complete the biophysical profile (BPP) for fetal well being | One day
  Assessment will done by determining fetal movement, fetal tone, fetal breathing, and amniotic fluid level

SECONDARY OUTCOMES:
Assess preliminary effectiveness and compare participant results to standard of care BPP | One day
  The results of BPP acquired with Pulsenmore device will be compared to standard of care BPP
Assess patient reported experience measures and patient reported outcomes with using the Pulsenmore home ultrasound device. | One day
  Patients will answer a questionnaire about their experience using Pulsenmore device

CONTACTS AND LOCATIONS:
Overall Officials: Alex Peahl, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No